CLINICAL TRIAL: NCT03772223
Title: A Phase 1, Randomized, Open-label, Single-dose, 3-way Cross-over Study to Compare the Pharmacokinetics of Budesonide and Albuterol Delivered by PT027 Compared With PT007 and PT008 Administered Separately (LOGAN).
Brief Title: A Study to Compare the Pharmacokinetics of Budesonide and Albuterol Delivered by PT027 Compared With PT007 and PT008 Administered Separately.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: D6930C00003
Record Dates: First submitted 2018-12-10; First posted 2018-12-11 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Healthy Volunteers
Keywords: Pharmacokinectics; Inhaled corticosteroid
MeSH Terms: interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Treatment sequence 1 (ABC) (Experimental): Participants will be randomized to each of the 6 different treatment sequences. Each treatment sequence consist of Treatment A (Budesonide/Albuterol Sulfate metered dose inhaler [BDA MDI] - PT027) , Treatment B (Budesonide metered dose inhaler [BD MDI] - PT008), and Treatment C (Albuterol Sulfate metered dose inhaler [AS MDI] - PT007). Each randomized participant will receive a single-dose (2 inhalations) on Day 1 of this Treatment Period.
  Interventions: Drug: Treatment A (Budesonide/Albuterol Sulfate metered dose inhaler); Drug: Treatment B (Budesonide metered dose inhaler); Drug: Treatment C (Albuterol Sulfate metered dose inhaler)
- Treatment sequence 2 (BCA) (Experimental): Participants will be randomized to each of the 6 different treatment sequences. Each treatment sequence consist of Treatment B (Budesonide metered dose inhaler [BD MDI] - PT008), Treatment C (Albuterol Sulfate metered dose inhaler [AS MDI] - PT007), and Treatment A (Budesonide/Albuterol Sulfate metered dose inhaler [BDA MDI] - PT027). Each randomized participant will receive a single-dose (2 inhalations) on Day 1 of this Treatment Period.
  Interventions: Drug: Treatment A (Budesonide/Albuterol Sulfate metered dose inhaler); Drug: Treatment B (Budesonide metered dose inhaler); Drug: Treatment C (Albuterol Sulfate metered dose inhaler)
- Treatment sequence 3 (CBA) (Experimental): Participants will be randomized to each of the 6 different treatment sequences. Each treatment sequence consist of Treatment C (Albuterol Sulfate metered dose inhaler [AS MDI] - PT007), Treatment B (Budesonide metered dose inhaler [BD MDI] - PT008), and Treatment A (Budesonide/Albuterol Sulfate metered dose inhaler [BDA MDI] - PT027). Each randomized participant will receive a single-dose (2 inhalations) on Day 1 of this Treatment Period.
  Interventions: Drug: Treatment A (Budesonide/Albuterol Sulfate metered dose inhaler); Drug: Treatment B (Budesonide metered dose inhaler); Drug: Treatment C (Albuterol Sulfate metered dose inhaler)
- Treatment sequence 4 (ACB) (Experimental): Participants will be randomized to each of the 6 different treatment sequences. Each treatment sequence consist of Treatment A (Budesonide/Albuterol Sulfate metered dose inhaler [BDA MDI] - PT027), Treatment C (Albuterol Sulfate metered dose inhaler [AS MDI] - PT007), and Treatment B (Budesonide metered dose inhaler [BD MDI] - PT008). Each randomized participant will receive a single-dose (2 inhalations) on Day 1 of this Treatment Period.
  Interventions: Drug: Treatment A (Budesonide/Albuterol Sulfate metered dose inhaler); Drug: Treatment B (Budesonide metered dose inhaler); Drug: Treatment C (Albuterol Sulfate metered dose inhaler)
- Treatment sequence 5 (BAC) (Experimental): Participants will be randomized to each of the 6 different treatment sequences. Each treatment sequence consist of Treatment B (Budesonide metered dose inhaler [BD MDI] - PT008), Treatment A (Budesonide/Albuterol Sulfate metered dose inhaler [BDA MDI] - PT027), and Treatment C (Albuterol Sulfate metered dose inhaler [AS MDI] - PT007). Each randomized participant will receive a single-dose (2 inhalations) on Day 1 of this Treatment Period.
  Interventions: Drug: Treatment A (Budesonide/Albuterol Sulfate metered dose inhaler); Drug: Treatment B (Budesonide metered dose inhaler); Drug: Treatment C (Albuterol Sulfate metered dose inhaler)
- Treatment sequence 6 (CAB) (Experimental): Participants will be randomized to each of the 6 different treatment sequences. Each treatment sequence consist of Treatment C (Albuterol Sulfate metered dose inhaler [AS MDI] - PT007), Treatment A (Budesonide/Albuterol Sulfate metered dose inhaler [BDA MDI] - PT027), and Treatment B (Budesonide metered dose inhaler [BD MDI] - PT008). Each randomized participant will receive a single-dose (2 inhalations) on Day 1 of this Treatment Period.
  Interventions: Drug: Treatment A (Budesonide/Albuterol Sulfate metered dose inhaler); Drug: Treatment B (Budesonide metered dose inhaler); Drug: Treatment C (Albuterol Sulfate metered dose inhaler)

INTERVENTIONS:
Drug: Treatment A (Budesonide/Albuterol Sulfate metered dose inhaler) — Randomized participants will receive a single-dose (2 inhalations, 2 x 80/90 µg).
Drug: Treatment B (Budesonide metered dose inhaler) — Randomized participants will receive a single-dose (2 inhalations, 2 x 80 µg).
Drug: Treatment C (Albuterol Sulfate metered dose inhaler) — Randomized participants will receive a single-dose (2 inhalations, 2 x 90 µg).

SUMMARY:
This is a Phase 1 study to compare the pharmacokinetics of budesonide and albuterol delivered by PT027 compared with PT007 and PT008 administered separately.

DETAILED DESCRIPTION:
This study will be a randomized, 3-way cross-over study in healthy male and female participants, performed at a single study centre. A total of 90 healthy male or female participants will be randomized in this study to ensure that at least 81 participants are evaluable.

The study will comprise:

A screening period of maximum 27 days; Three treatment periods during which participants will be resident from the morning before dosing with Budesonide/Albuterol Sulfate metered dose inhaler (BDA MDI), Budesonide metered dose inhaler (BD MDI), and Albuterol Sulfate metered dose inhaler (AS MDI [Day -1]) until at least 24 hours after dosing; discharged on the morning of Day 2; and A final visit within 5 to 7 days after the last administration of BDA MDI, BD MDI, or AS MDI.

There will be a minimum washout period of 7 days between each dose administration.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures.
2. Healthy male and female participants aged 18 to 55 years (inclusive) with suitable veins for cannulation or repeated venipuncture.
3. Females must have a negative pregnancy test at the Screening Visit and on admission to the Clinical Unit and must not be lactating.
4. Have a body mass index between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.
5. Must be able to demonstrate proper inhalation technique using the AIM device and placebo MDI at the Screening Visit.
6. Forced expiratory volume in 1 second in litres (FEV1) ≥ 80% of predicted value and forced vital capacity in litres (FEV1)/FVC ratio ≥ 70%.

Exclusion Criteria:

1. Pregnant or nursing female participants or participants who are trying to conceive.
2. For female participants, a positive serum human chorionic gonadotropin (hCG) test at screening or a positive urine hCG at admission for any of the 3 Treatment Periods.
3. History of any clinically significant disease or disorder which, in the opinion of the Principal Investigator (PI), may either put the subject at risk because of participation in the study, or influence the results or the participant's ability to participate in the study.
4. History or presence of gastrointestinal, hepatic or renal disease, or any other condition known to interfere with absorption, distribution, metabolism, or excretion of drugs.
5. Participants who have cancer that has not been in complete remission for at least 5 years.
6. Any history of asthma or Chronic obstructive pulmonary disease.
7. Any clinically significant illness, medical/surgical procedure, or trauma within 4 weeks of the first administration of Investigational Medicinal Product (IMP).
8. Any clinically significant abnormalities in clinical chemistry, haematology, or urinalysis results, at the Screening Visit as judged by the PI.
9. Any clinically significant abnormal findings in vital signs at the Screening Visit, as judged by the PI.
10. Any clinically significant abnormalities on 12-lead electrocardiogram at the Screening Visit, as judged by the PI.
11. Any positive result on screening for serum hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus antibody.
12. Known or suspected history of drug abuse in the past 2 years, as judged by the PI.
13. Has received another new chemical entity (defined as a compound which has not been approved for marketing) within 3 months of the first administration of IMP in this study. The period of exclusion begins 3 months after the final dose or 1 month after the last visit whichever is the longest.
14. Plasma donation within 1 month of screening or any blood donation/loss more than 500 mL during the 3 months prior to screening.
15. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the PI or history of hypersensitivity to drugs with a similar chemical structure or class to budesonide and albuterol sulfate.
16. Current smokers or those who have smoked or used nicotine products (including e cigarettes) within the 3 months prior to screening.
17. Positive screen for drugs of abuse, cotinine or alcohol at the Screening Visit or on each admission to the Clinical Unit.
18. Use of drugs with enzyme-inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.
19. Use of any prescribed or non prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of IMP or longer if the medication has a long half life.
20. Known or suspected history of alcohol or excessive intake of alcohol in the last 2 years as judged by the PI.
21. Involvement of any AstraZeneca, PAREXEL or study site employee or their close relatives.
22. Judgment by the PI that the participant should not participate in the study if they have any ongoing or recent (i.e., during the screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions, and requirements.
23. Vulnerable participant, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-10 (Actual)

PRIMARY OUTCOMES:
AUC for albuterol | At Day 1 (pre-dose and 5, 15, 20, 30 and 45 minutes and 1, 2, 3, 4, 6, 8, 10 and 12 hours post dose), and Day 2 (24 hours post dose)
  To determine the area under the plasma concentration-time curve from time zero to infinity (AUC) after single dose administration of albuterol delivered via BDA MDI with BD MDI monotherapy and AS MDI monotherapy.
AUC for budesonide | At Day 1 (pre-dose and 5, 15, 20, 30 and 45 minutes and 1, 2, 3, 4, 6, 8, 10 and 12 hours post dose), and Day 2 (24 hours post dose)
  To determine the AUC after single dose administration of budesonide delivered via BDA MDI with BD MDI monotherapy and AS MDI monotherapy.
AUC(0-t) for albuterol | At Day 1 (pre-dose and 5, 15, 20, 30 and 45 minutes and 1, 2, 3, 4, 6, 8, 10 and 12 hours post dose), and Day 2 (24 hours post dose)
  To determine the area under the plasma concentration time curve from time zero to time of last quantifiable concentration (AUC([0-t]) after single dose administration of albuterol delivered via BDA MDI with BD MDI monotherapy and AS MDI monotherapy.
AUC(0-t) for budesonide | At Day 1 (pre-dose and 5, 15, 20, 30 and 45 minutes and 1, 2, 3, 4, 6, 8, 10 and 12 hours post dose), and Day 2 (24 hours post dose)
  To determine the AUC(0-t) after single dose administration of budesonide delivered via BDA MDI with BD MDI monotherapy and AS MDI monotherapy.
Cmax for albuterol | At Day 1 (pre-dose and 5, 15, 20, 30 and 45 minutes and 1, 2, 3, 4, 6, 8, 10 and 12 hours post dose), and Day 2 (24 hours post dose)
  To determine observed maximum plasma concentration (Cmax) after single dose administration of albuterol delivered via BDA MDI with BD MDI monotherapy and AS MDI monotherapy.
Cmax for budesonide | At Day 1 (pre-dose and 5, 15, 20, 30 and 45 minutes and 1, 2, 3, 4, 6, 8, 10 and 12 hours post dose), and Day 2 (24 hours post dose)
  To determine Cmax after single dose administration of budesonide delivered via BDA MDI with BD MDI monotherapy and AS MDI monotherapy.

SECONDARY OUTCOMES:
tlast for albuterol | At Day 1 (pre-dose and 5, 15, 20, 30 and 45 minutes and 1, 2, 3, 4, 6, 8, 10 and 12 hours post dose), and Day 2 (24 hours post dose)
  To determine the time of last quantifiable plasma concentration (tlast) after single dose administration of albuterol delivered via BDA MDI with BD MDI monotherapy and AS MDI monotherapy.
tlast for budesonide | At Day 1 (pre-dose and 5, 15, 20, 30 and 45 minutes and 1, 2, 3, 4, 6, 8, 10 and 12 hours post dose), and Day 2 (24 hours post dose)
  To determine the tlast after single dose administration of budesonide delivered via BDA MDI with BD MDI monotherapy and AS MDI monotherapy.
tmax for albuterol | At Day 1 (pre-dose and 5, 15, 20, 30 and 45 minutes and 1, 2, 3, 4, 6, 8, 10 and 12 hours post dose), and Day 2 (24 hours post dose)
  To determine time to reach maximum observed plasma concentration (tmax) after single dose administration of albuterol delivered via BDA MDI with BD MDI monotherapy and AS MDI monotherapy.
tmax for budesonide | At Day 1 (pre-dose and 5, 15, 20, 30 and 45 minutes and 1, 2, 3, 4, 6, 8, 10 and 12 hours post dose), and Day 2 (24 hours post dose)
  To determine tmax after single dose administration of budesonide delivered via BDA MDI with BD MDI monotherapy and AS MDI monotherapy.
t1/2λz for albuterol | At Day 1 (pre-dose and 5, 15, 20, 30 and 45 minutes and 1, 2, 3, 4, 6, 8, 10 and 12 hours post dose), and Day 2 (24 hours post dose)
  To determine the time to apparent elimination half-life (t1/2λz)after single dose administration of albuterol delivered via BDA MDI with BD MDI monotherapy and AS MDI monotherapy
t1/2λz for budesonide | At Day 1 (pre-dose and 5, 15, 20, 30 and 45 minutes and 1, 2, 3, 4, 6, 8, 10 and 12 hours post dose), and Day 2 (24 hours post dose)
  To determine t1/2λz after single dose administration of budesonide delivered via BDA MDI with BD MDI monotherapy and AS MDI monotherapy.
λz for albuterol | At Day 1 (pre-dose and 5, 15, 20, 30 and 45 minutes and 1, 2, 3, 4, 6, 8, 10 and 12 hours post dose), and Day 2 (24 hours post dose)
  To determine the terminal elimination rate constant (λz) after single dose administration of albuterol delivered via BDA MDI with BD MDI monotherapy and AS MDI monotherapy.
λz for budesonide | At Day 1 (pre-dose and 5, 15, 20, 30 and 45 minutes and 1, 2, 3, 4, 6, 8, 10 and 12 hours post dose), and Day 2 (24 hours post dose)
  To determine the λz after single dose administration of budesonide delivered via BDA MDI with BD MDI monotherapy and AS MDI monotherapy.
CL/F for albuterol | At Day 1 (pre-dose and 5, 15, 20, 30 and 45 minutes and 1, 2, 3, 4, 6, 8, 10 and 12 hours post dose), and Day 2 (24 hours post dose)
  To determine the apparent total body clearance of drug from plasma after extravascular administration (CL/F) after single dose administration of albuterol delivered via BDA MDI with BD MDI monotherapy and AS MDI monotherapy.
CL/F for budesonide | At Day 1 (pre-dose and 5, 15, 20, 30 and 45 minutes and 1, 2, 3, 4, 6, 8, 10 and 12 hours post dose), and Day 2 (24 hours post dose)
  To determine the CL/F after single dose administration of budesonide delivered via BDA MDI with BD MDI monotherapy and AS MDI monotherapy.
Vz/F for albuterol | At Day 1 (pre-dose and 5, 15, 20, 30 and 45 minutes and 1, 2, 3, 4, 6, 8, 10 and 12 hours post dose), and Day 2 (24 hours post dose)
  To determine the apparent volume of distribution during the terminal phase after extravascular administration (Vz/F) after single dose administration of albuterol delivered via BDA MDI with BD MDI monotherapy and AS MDI monotherapy.
Vz/F for budesonide | At Day 1 (pre-dose and 5, 15, 20, 30 and 45 minutes and 1, 2, 3, 4, 6, 8, 10 and 12 hours post dose), and Day 2 (24 hours post dose)
  To determine the Vz/F after single dose administration of budesonide delivered via BDA MDI with BD MDI monotherapy and AS MDI monotherapy.
Number of participants with adverse events (AEs)/serious AEs (SAEs) | From Screening to Post-study Visit (5-7 days)
  To assess the safety and tolerability of BDA MDI, BD MDI, and AS MDI.

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Forte Soto, Principal Investigator — Parexel
Locations (1):
- Research Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided